CLINICAL TRIAL: NCT02057939
Title: Salvage Therapeutic Radiation With Enzalutamide and ADT in Men With Recurrent Prostate Cancer (STREAM)
Acronym: STREAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medivation, Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00049865
Record Dates: First submitted 2014-01-31; First posted 2014-02-07 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; enzalutamide; ADT; radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzalutamide (Experimental): Enzalutamide, Androgen Deprivation, and Radiation Therapy
  Interventions: Drug: enzalutamide; Drug: Androgen Deprivation; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: enzalutamide — 160 mg orally once daily for six months
  Other Names: Xtandi
Drug: Androgen Deprivation — Two injections each lasting three months, for a total of six months of androgen deprivation therapy. Doctor will help determine which androgen deprivation drug to use.
  Other Names: leuprolide acetate (Lupron Depot, 22.5 mg)
Radiation: Radiation Therapy — Daily (Monday-Friday) for 6-8 weeks, final dose of approximately 66 Gy

SUMMARY:
The purpose of this study is to describe the 2 year progression-free survival in men with recurrent PSA-only disease after prostatectomy receiving combined enzalutamide and standard androgen-deprivation therapy (ADT) with salvage radiation therapy. Eligible men will have recurrent PSA-only prostate cancer within 4 years of prostatectomy, and a PSA of 0.2 - 4 in the absence of metastatic disease on CT and bone scans. In addition to standard ADT and radiation therapy, research participants will take enzalutamide once daily for six months. It is primarily hypothesized the 2 year PFS rate will be improved with the combined therapy compared to the historical control data in a similar patients setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma. Variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate, are not permitted.
* Gleason sum of 7, 8, 9, or 10 at the time of prostatectomy.
* PSA relapse within 4 years of prostatectomy defined by persistently detectable or rising PSA after surgery.
* Evidence of disease recurrence or progression as evidenced by a PSA > 0.20. This requires 2 consecutive rises in PSA, at least 1 week apart, over the post-prostatectomy nadir or one PSA value above 0.20 ng/mL if the patient failed to achieve a post-prostatectomy nadir of < 0.2 ng/mL.
* Age ≥ 18 years
* Karnofsky performance status ≥ 70
* Adequate laboratory parameters
* Adequate bone marrow function: ANC ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hb >9g/dL
* AST/SGOT and ALT/SGPT ≤ 2.5 x Institutional Upper Limit of Normal (ULN)
* Serum bilirubin ≤ 1.5 x Institutional ULN
* Serum creatinine ≤ 1.5 x Institutional ULN or 24-hour clearance ≥ 50 mL/min
* A minimum of 4 weeks from any major surgery prior to registration.
* Ability to swallow, retain, and absorb oral medication.
* Ability to understand and the willingness to sign a written informed consent document.
* Must use a condom if having sex with a pregnant woman.
* Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration.

Exclusion Criteria:

* Radiographic evidence of metastatic disease. Patients with node-positive disease (<2 positive nodes) at the time of radical prostatectomy are eligible. Patients with pelvic nodes up to 2 cm by short axis at the time of screening are eligible. Patients with any enlarged lymph nodes in the retroperitoneum or above the aortic bifurcation or with pelvic nodes ≥ 2 cm must be excluded.
* PSA > 4.0 ng/mL.
* Testosterone level ≤ 100 ng/dL.
* More than 1 month of prior hormone exposure or hormone exposure within 30 days of registration. Prior enzalutamide, ketoconazole, abiraterone, or TAK700 prohibited. Prior 5α reductase inhibitors are allowed.
* Prior immunotherapy including sipuleucel-T.
* Prior systemic chemotherapy (docetaxel, cabazitaxel, estramustine, other cytotoxic agents)
* History of solid organ or stem cell transplantation.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, prior head or traumatic brain injury with loss of consciousness, prior or current space-occupying lesion in the brain). Also, history of loss of consciousness or transient ischemic attack within 12 months of Day 1 visit.
* Known or suspected brain metastasis or active leptomeningeal disease.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of enzalutamide or increase the risk of radiation (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndromes, prior small bowel resection, or inflammatory bowel disease).
* Patients who have received prior prostate or pelvic radiotherapy, including external beam or brachytherapy.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy prior to registration.
* Patients unable or unwilling to abide by the study protocol or cooperate fully with the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD ScM FACP, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Bitting RL, Healy P, George DJ, Anand M, Kim S, Mayer T, Winters C, Riggan C, Rasmussen J, Wilder R, Stein M, Frizzell B, Harrison MR, Zhang T, Lee WR, Wu Y, Koontz BF, Armstrong AJ. Phase II Trial of Enzalutamide and Androgen Deprivation Therapy with Salvage Radiation in Men with High-risk Prostate-specific Antigen Recurrent Prostate Cancer: The STREAM Trial. Eur Urol Oncol. 2021 Dec;4(6):948-954. doi: 10.1016/j.euo.2020.01.005. Epub 2020 Feb 13. PMID 32063492

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enzalutamide
Started | 38
Completed | 37
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Two Year Progression-free Survival
Description: Percentage of patients surviving 2 years from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of first documented progression or death due to any cause. Progression-free was defined as being without one of the following: serum PSA value of 0.2 ng/mL or more above post-radiotherapy PSA nadir that continues to increase 4 weeks later OR if no nadir is experienced, two rising PSA values over 4 or more weeks OR evidence of clinical progression or initiation of systemic therapy for progressive disease
Time Frame: 2 years
Population: One patient did not receive radiotherapy due to continual scar tissue development surrounding the ureters. This patient is not considered for analyses.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
percentage | 64.9 [47.3 to 77.9]

2. Secondary Outcome: PSA Less Than 0.1
Description: The percentage of men with PSA less than 0.1 ng/mL and testosterone greater than 100
Time Frame: every year, up to 3 years
Population: One patient did not receive radiotherapy due to continual scar tissue development surrounding the ureters. This patient is not considered for analyses. Note that 11 patients did not have PSA measurements at 2 years and 24 did not have PSA measurements at 3 years. They are still included in the denominator.
Measure: Number; unit: percentage
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
percentage
  1 year | 75.7
  2 year | 48.6
  3 year | 32.4

3. Secondary Outcome: Three Year Progression-free Survival
Description: Percentage of patients surviving 3 years from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of first documented progression or death due to any cause. Progression-free was defined as being without one of the following: serum PSA value of 0.2 ng/mL or more above post-radiotherapy PSA nadir that continues to increase 4 weeks later OR if no nadir is experienced, two rising PSA values over 4 or more weeks OR evidence of clinical progression or initiation of systemic therapy for progressive disease
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
percentage | 53.2 [35.9 to 67.9]

4. Secondary Outcome: Biochemical Progression-free Survival
Description: Percentage of patients surviving 2 and 3 years from the start of study treatment without progression of disease. Biochemical PFS was defined as the time from the date of study treatment initiation to the date of first documented progression or death due to any cause. Progression-free was defined as being without one of the following: serum PSA value of 0.2 ng/mL or more above post-radiotherapy PSA nadir that continues to increase 4 weeks later OR if no nadir is experienced, two rising PSA values over 4 or more weeks
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
percentage
  2 year bPFS | 64.9 [47.3 to 77.9]
  3 year bPFS | 53.2 [35.9 to 67.9]

5. Secondary Outcome: PSA Nadir
Description: Median PSA nadir post-radiation therapy
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
ng/ml | 0 [0 to 0.1]

6. Secondary Outcome: Time to Testosterone Recovery
Description: Percentage of patients with recovering testosterone to > 100 at 1, 2, and 3 years.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Enzalutamide
Number analyzed (Participants) | 37
percentage
  1 year | 94.6
  2 year | 100
  3 year | 100

7. Secondary Outcome: Number of Patients With Adverse Events Related to Combination Enzalutamide, ADT, and XRT
Description: Safety and tolerability will be assessed using CTCAE v4.0
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 38
participants | 36

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=38)
Myocardial infarction (Cardiac disorders) | 1
Other, Specify: BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=38)
Anemia (Blood and lymphatic system disorders) | 9
Acute coronary syndrome (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Other, Specify: EAR PRESSURE (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Other, Specify: FLOATERS (Eye disorders) | 1
Other, Specify: PSUEDOPHAKIA (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 30
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
Injection site reaction (General disorders) | 1
Irritability (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 6
Bronchial infection (Infections and infestations) | 1
Other, Specify: COMMON COLD (Infections and infestations) | 1
Other, Specify: TICK BITE WITH FEVER, CHILLS, BODY ACHES, HEADACHES (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Skin infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 1
Weight gain (Investigations) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Other, Specify (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Akathisia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 7
Memory impairment (Nervous system disorders) | 5
Movements involuntary (Nervous system disorders) | 1
Other, Specify: RESTLESS LEG SYNDROME (Nervous system disorders) | 1
Other, Specify: RESTLESS LEGS (Nervous system disorders) | 5
Other, Specify: RESTLESS LEGS; INTERMITTENT/AT NIGHT (Nervous system disorders) | 1
Other, Specify: VIVID DREAMS (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 15
Libido decreased (Psychiatric disorders) | 3
Personality change (Psychiatric disorders) | 2
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Other, Specify: NOCTURIA (Renal and urinary disorders) | 2
Other, Specify: NOCTURIA, RELATED TO RADIATION (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 11
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 4
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 5
Breast pain (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Other, Specify: A LUMP JUST ABOVE ANTECUBITAL SPACE OF LEFT ARM (Skin and subcutaneous tissue disorders) | 1
Other, Specify: ABRASION WITH EDEMA, LEFT ANKLE, DUE TO TRAUMA TO LEFT LEG (Skin and subcutaneous tissue disorders) | 1
Other, Specify: ECZEMA BILATERAL ELBOWS AND LEFT SHIN (Skin and subcutaneous tissue disorders) | 1
Other, Specify: ONE SPOT ON EACH ARM (Skin and subcutaneous tissue disorders) | 1
Other, Specify: SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Other, Specify: MOHS SURGERY FOR BASAL CELL (Surgical and medical procedures) | 1
Other, Specify: RECTAL IRRITATION, RELATED TO RADIATION (Surgical and medical procedures) | 1
Hot flashes (Vascular disorders) | 28
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02057939/Prot_SAP_000.pdf